CLINICAL TRIAL: NCT01991353
Title: Prospective, Double Blind, Randomized Trial: Meniscal Repair With or Without Augmentation Utilizing Platelet Rich Plasma.
Brief Title: Platelet Rich Plasma Study With Meniscal Repair
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Fraser Orthopaedic Research Society (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-122
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Meniscus Lesion
Keywords: Knee; meniscus; platelet rich plasma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- With PRP (Experimental): Standardized meniscal repair with PRP (platelet rich plasma) in the meniscal healing bed.
  Interventions: Procedure: With PRP
- Without PRP (Active Comparator): Standardized meniscal repair without PRP (platelet rich plasma).
  Interventions: Procedure: Without PRP

INTERVENTIONS:
Procedure: With PRP — Following meniscal repair, PRFM will be delivered arthroscopically into the tear site using a portal skid, arthroscopic canula and arthroscopic atraumatic tissue grasper into the interface of the repair site.
  Other Names: Platelet Rich Fibrin Matrix (PRFM)
  Arms: With PRP
Procedure: Without PRP — Standard of care meniscal repair without augmentation.
  Arms: Without PRP

SUMMARY:
This study will compare meniscal healing with or without platelet rich plasma. The assessments will include validated, disease specific, patient oriented outcome measures, MRI arthrogram (MRA). Results of this study will help ascertain whether PRP improves meniscal healing rates.

Null Hypothesis: There is no difference in meniscal healing with or without the use of PRP.

DETAILED DESCRIPTION:
The integrity of the meniscus is pivotal to the distribution of joint reaction forces and shock absorption across the knee and meniscal damage can lead to secondary degenerative joint disease. This has lead to treatments directed towards repairing and preserving the meniscus to alter the progression of joint degeneration. Although success rates of meniscal repair are greater when performed in association with anterior cruciate reconstruction, healing rates remain in the 70-80% range for isolated repairs.

Therefore, techniques such as the use of fibrin clots, trephining and rasping of the tissues, have been incorporated to improve healing results of meniscal repair. There has been a surge of enthusiasm for the use of Platelet Rich Plasma (PRP) to improve healing rates of soft tissue injuries. Therefore, it may be reasonable to surmise that applying blood products, such as thrombin and platelet rich plasma, to the meniscal repair bed may induce more complete and possibly faster healing.

ELIGIBILITY:
Inclusion Criteria:

* complete vertical longitudinal tear > 10 mm in length
* tear located in the vascular portion of the meniscus, classified as either red-red or red-white zones
* a stable knee, or a knee that is stabilized with a concurrent ACL reconstruction
* unstable peripheral tear that can be displaced toward center of joint
* single tear of the medial and/or lateral meniscus
* skeletally mature patients 18-60 years of age

Exclusion Criteria:

* associated significant ligament instability: Grade III MCL, Grade III PCL
* discoid meniscus
* ACL deficient knee
* Outerbridge Grade III or IV cartilage changes on arthroscopy in the involved compartment
* Significant degenerative changes on radiographs (Kellgren Lawrence >/= Grade III)
* Associated osteochondral defect that requires treatment
* Inflammatory arthropathy (e.g. rheumatoid arthritis)
* Non repairable meniscus (ie white zone, irreducible meniscus)
* Degenerative meniscus or presence of CPP crystals in meniscus
* Underlying bleeding disorder or coagulopathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2017-07 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
MRA (magnetic resonance imaging arthrography | 6 months
  The primary outcome measures will be assessment of meniscal healing integrity using magnetic resonance imaging arthrography six months post repair.

SECONDARY OUTCOMES:
WOMET - Western Ontario Meniscal Outcome Measure | Baseline, 3 months, 6 months 12 months
  The WOMET is a disease-specific validated tool designed to evaluate HRQOL (Health Related Quality of Life) in patients with meniscal pathology (meniscal tears or in patients who have undergone meniscal repair or resection). In this subset of patients with meniscal pathology, the WOMET has been found to be reliable, valid and responsive.
  The WOMET has 16 items including the domains of physical symptoms, sports/recreation/work/lifestyle, and emotions. It demonstrated adequate content and construct validity when compared with other measures. Test-retest reliability was assessed and was found to be high, with an intraclass correlation coefficient of 0.833.
VAS Pain Score - Visual Analog Scale | Baseline, Post-op Day 1, 6 weeks
  Pain Visual Analog Scale.
Range of motion | 6 weeks, 3 months, 6 months, 12 months
  Knee range of motion measurements.
Tegner Score | Baseline, 3, 6 and 12 months post treatment
  Return to pre injury activity level as measured by the Tegner Score.

OTHER OUTCOMES:
Second look arthroscopy | if applicable
  If a second look arthroscopy is performed, the status of the meniscus (healed or not healed) will be compared to the MRA findings. Second look arthroscopy will be performed on subjects with clinical indication of a failed meniscal repair. Clinical indications of failed meniscus repair include persistent pain and symptoms or MRA positive for a meniscus repair.

CONTACTS AND LOCATIONS:
Overall Officials: Robert G. McCormack, MD, FRCSC, Principal Investigator — Simon Fraser Orthopaedic Fund / Fraser Health Authority / University of British Columbia
Locations (1):
- Eagle Ridge Hospital, Port Moody, British Columbia, Canada

REFERENCES:
- [Result] Andersson-Molina H, Karlsson H, Rockborn P. Arthroscopic partial and total meniscectomy: A long-term follow-up study with matched controls. Arthroscopy. 2002 Feb;18(2):183-9. doi: 10.1053/jars.2002.30435. PMID 11830813
- [Result] Johnson RJ, Kettelkamp DB, Clark W, Leaverton P. Factors effecting late results after meniscectomy. J Bone Joint Surg Am. 1974 Jun;56(4):719-29. No abstract available. PMID 4406907
- [Result] Greis PE, Holmstrom MC, Bardana DD, Burks RT. Meniscal injury: II. Management. J Am Acad Orthop Surg. 2002 May-Jun;10(3):177-87. doi: 10.5435/00124635-200205000-00004. PMID 12041939
- [Result] Lietman SA, Hobbs W, Inoue N, Reddi AH. Effects of selected growth factors on porcine meniscus in chemically defined medium. Orthopedics. 2003 Aug;26(8):799-803. doi: 10.3928/0147-7447-20030801-19. PMID 12938945
- [Result] Sethi PM, Cooper A, Jokl P. Technical tips in orthopaedics: meniscal repair with use of an in situ fibrin clot. Arthroscopy. 2003 May-Jun;19(5):E44. doi: 10.1053/jars.2003.50164. PMID 12724668
- [Result] Henning CE, Lynch MA, Yearout KM, Vequist SW, Stallbaumer RJ, Decker KA. Arthroscopic meniscal repair using an exogenous fibrin clot. Clin Orthop Relat Res. 1990 Mar;(252):64-72. PMID 2406075
- [Result] Henning CE, Yearout KM, Vequist SW, Stallbaumer RJ, Decker KA. Use of the fascia sheath coverage and exogenous fibrin clot in the treatment of complex meniscal tears. Am J Sports Med. 1991 Nov-Dec;19(6):626-31. doi: 10.1177/036354659101900613. PMID 1781502
- [Result] van Trommel MF, Simonian PT, Potter HG, Wickiewicz TL. Arthroscopic meniscal repair with fibrin clot of complete radial tears of the lateral meniscus in the avascular zone. Arthroscopy. 1998 May-Jun;14(4):360-5. doi: 10.1016/s0749-8063(98)70002-7. PMID 9620646
- [Result] Voloshin AS, Wosk J. Shock absorption of meniscectomized and painful knees: a comparative in vivo study. J Biomed Eng. 1983 Apr;5(2):157-61. doi: 10.1016/0141-5425(83)90036-5. PMID 6687914
- [Result] Walker PS, Erkman MJ. The role of the menisci in force transmission across the knee. Clin Orthop Relat Res. 1975;(109):184-92. doi: 10.1097/00003086-197506000-00027. PMID 1173360
- [Result] Kettelkamp DB, Jacobs AW. Tibiofemoral contact area--determination and implications. J Bone Joint Surg Am. 1972 Mar;54(2):349-56. No abstract available. PMID 4678847
- [Result] Fukubayashi T, Kurosawa H. The contact area and pressure distribution pattern of the knee. A study of normal and osteoarthrotic knee joints. Acta Orthop Scand. 1980 Dec;51(6):871-9. doi: 10.3109/17453678008990887. PMID 6894212
- [Result] Cox JS, Nye CE, Schaefer WW, Woodstein IJ. The degenerative effects of partial and total resection of the medial meniscus in dogs' knees. Clin Orthop Relat Res. 1975;(109):178-83. doi: 10.1097/00003086-197506000-00026. PMID 1173359
- [Result] Rangger C, Klestil T, Gloetzer W, Kemmler G, Benedetto KP. Osteoarthritis after arthroscopic partial meniscectomy. Am J Sports Med. 1995 Mar-Apr;23(2):240-4. doi: 10.1177/036354659502300219. PMID 7778712
- [Result] McDermott ID, Amis AA. The consequences of meniscectomy. J Bone Joint Surg Br. 2006 Dec;88(12):1549-56. doi: 10.1302/0301-620X.88B12.18140. PMID 17159163
- [Result] FAIRBANK TJ. Knee joint changes after meniscectomy. J Bone Joint Surg Br. 1948 Nov;30B(4):664-70. No abstract available. PMID 18894618
- [Result] Fauno P, Nielsen AB. Arthroscopic partial meniscectomy: a long-term follow-up. Arthroscopy. 1992;8(3):345-9. doi: 10.1016/0749-8063(92)90066-k. PMID 1418207
- [Result] DeHaven KE, Black KP, Griffiths HJ. Open meniscus repair. Technique and two to nine year results. Am J Sports Med. 1989 Nov-Dec;17(6):788-95. doi: 10.1177/036354658901700612. PMID 2696377
- [Result] DeHaven KE. Meniscus repair. Am J Sports Med. 1999 Mar-Apr;27(2):242-50. doi: 10.1177/03635465990270022301. No abstract available. PMID 10102109
- [Result] DeHaven KE, Lohrer WA, Lovelock JE. Long-term results of open meniscal repair. Am J Sports Med. 1995 Sep-Oct;23(5):524-30. doi: 10.1177/036354659502300502. PMID 8526265
- [Result] Rodeo SA. Arthroscopic meniscal repair with use of the outside-in technique. Instr Course Lect. 2000;49:195-206. PMID 10829175
- [Result] Toman CV, Dunn WR, Spindler KP, Amendola A, Andrish JT, Bergfeld JA, Flanigan D, Jones MH, Kaeding CC, Marx RG, Matava MJ, McCarty EC, Parker RD, Wolcott M, Vidal A, Wolf BR, Huston LJ, Harrell FE Jr, Wright RW. Success of meniscal repair at anterior cruciate ligament reconstruction. Am J Sports Med. 2009 Jun;37(6):1111-5. doi: 10.1177/0363546509337010. PMID 19465734
- [Result] Horibe S, Shino K, Nakata K, Maeda A, Nakamura N, Matsumoto N. Second-look arthroscopy after meniscal repair. Review of 132 menisci repaired by an arthroscopic inside-out technique. J Bone Joint Surg Br. 1995 Mar;77(2):245-9. PMID 7706339
- [Result] Horibe S, Shino K, Maeda A, Nakamura N, Matsumoto N, Ochi T. Results of isolated meniscal repair evaluated by second-look arthroscopy. Arthroscopy. 1996 Apr;12(2):150-5. doi: 10.1016/s0749-8063(96)90003-1. PMID 8776990
- [Result] Logan M, Watts M, Owen J, Myers P. Meniscal repair in the elite athlete: results of 45 repairs with a minimum 5-year follow-up. Am J Sports Med. 2009 Jun;37(6):1131-4. doi: 10.1177/0363546508330138. Epub 2009 Mar 11. PMID 19279222
- [Result] White LM, Schweitzer ME, Weishaupt D, Kramer J, Davis A, Marks PH. Diagnosis of recurrent meniscal tears: prospective evaluation of conventional MR imaging, indirect MR arthrography, and direct MR arthrography. Radiology. 2002 Feb;222(2):421-9. doi: 10.1148/radiol.2222010396. PMID 11818609
- [Result] Ciliz D, Ciliz A, Elverici E, Sakman B, Yuksel E, Akbulut O. Evaluation of postoperative menisci with MR arthrography and routine conventional MRI. Clin Imaging. 2008 May-Jun;32(3):212-9. doi: 10.1016/j.clinimag.2007.09.008. PMID 18502349
- [Result] Vives MJ, Homesley D, Ciccotti MG, Schweitzer ME. Evaluation of recurring meniscal tears with gadolinium-enhanced magnetic resonance imaging: a randomized, prospective study. Am J Sports Med. 2003 Nov-Dec;31(6):868-73. doi: 10.1177/03635465030310062301. PMID 14623651
- [Result] Elentuck D, Palmer WE. Direct magnetic resonance arthrography. Eur Radiol. 2004 Nov;14(11):1956-67. doi: 10.1007/s00330-004-2449-3. Epub 2004 Sep 3. PMID 15351900
- [Result] Schulte-Altedorneburg G, Gebhard M, Wohlgemuth WA, Fischer W, Zentner J, Wegener R, Balzer T, Bohndorf K. MR arthrography: pharmacology, efficacy and safety in clinical trials. Skeletal Radiol. 2003 Jan;32(1):1-12. doi: 10.1007/s00256-002-0595-8. Epub 2002 Dec 5. PMID 12525938
- [Result] Quinn SF, Brown TF. Meniscal tears diagnosed with MR imaging versus arthroscopy: how reliable a standard is arthroscopy? Radiology. 1991 Dec;181(3):843-7. doi: 10.1148/radiology.181.3.1947108.
- [Result] Deutsch AL, Mink JH, Fox JM, Arnoczky SP, Rothman BJ, Stoller DW, Cannon WD Jr. Peripheral meniscal tears: MR findings after conservative treatment or arthroscopic repair. Radiology. 1990 Aug;176(2):485-8. doi: 10.1148/radiology.176.2.2367665.
- [Result] De Smet AA, Norris MA, Yandow DR, Quintana FA, Graf BK, Keene JS. MR diagnosis of meniscal tears of the knee: importance of high signal in the meniscus that extends to the surface. AJR Am J Roentgenol. 1993 Jul;161(1):101-7. doi: 10.2214/ajr.161.1.8517286.
- [Result] Haims AH, Katz LD, Ruwe PA. MR Arthrography of the Knee. Semin Musculoskelet Radiol. 1998;2(4):385-396. doi: 10.1055/s-2008-1080119. PMID 11387117
- [Result] Cardello P, Gigli C, Ricci A, Chiatti L, Voglino N, Pofi E. Retears of postoperative knee meniscus: findings on magnetic resonance imaging (MRI) and magnetic resonance arthrography (MRA) by using low and high field magnets. Skeletal Radiol. 2009 Feb;38(2):149-56. doi: 10.1007/s00256-008-0600-y. Epub 2008 Oct 10. PMID 18846372
- [Result] Gopez AG, Kavanagh EC. MR imaging of the postoperative meniscus: repair, resection, and replacement. Semin Musculoskelet Radiol. 2006 Sep;10(3):229-40. doi: 10.1055/s-2006-957176. PMID 17195131
- [Result] Muellner T, Egkher A, Nikolic A, Funovics M, Metz V. Open meniscal repair: clinical and magnetic resonance imaging findings after twelve years. Am J Sports Med. 1999 Jan-Feb;27(1):16-20. doi: 10.1177/03635465990270011001. PMID 9934413
- [Result] White LM, Kramer J, Recht MP. MR imaging evaluation of the postoperative knee: ligaments, menisci, and articular cartilage. Skeletal Radiol. 2005 Aug;34(8):431-52. doi: 10.1007/s00256-005-0914-y. Epub 2005 Jun 21. PMID 15968555
- [Result] Mustonen AO, Tielinen L, Lindahl J, Hirvensalo E, Kiuru M, Koskinen SK. MRI of menisci repaired with bioabsorbable arrows. Skeletal Radiol. 2006 Jul;35(7):515-21. doi: 10.1007/s00256-006-0080-x. Epub 2006 Mar 18. PMID 16547748
- [Result] Scott GA, Jolly BL, Henning CE. Combined posterior incision and arthroscopic intra-articular repair of the meniscus. An examination of factors affecting healing. J Bone Joint Surg Am. 1986 Jul;68(6):847-61. PMID 3755440
- [Result] Arnoczky SP, Cooper TG, Stadelmaier DM, Hannafin JA. Magnetic resonance signals in healing menisci: an experimental study in dogs. Arthroscopy. 1994 Oct;10(5):552-7. doi: 10.1016/s0749-8063(05)80013-1. PMID 7999166
- [Result] Arnoczky SP, Warren RF. The microvasculature of the meniscus and its response to injury. An experimental study in the dog. Am J Sports Med. 1983 May-Jun;11(3):131-41. doi: 10.1177/036354658301100305. PMID 6688156
- [Result] Applegate GR, Flannigan BD, Tolin BS, Fox JM, Del Pizzo W. MR diagnosis of recurrent tears in the knee: value of intraarticular contrast material. AJR Am J Roentgenol. 1993 Oct;161(4):821-5. doi: 10.2214/ajr.161.4.8372768.
- [Result] Wojtys EM, Chan DB. Meniscus structure and function. Instr Course Lect. 2005;54:323-30. PMID 15948460
- [Result] Hashimoto J, Kurosaka M, Yoshiya S, Hirohata K. Meniscal repair using fibrin sealant and endothelial cell growth factor. An experimental study in dogs. Am J Sports Med. 1992 Sep-Oct;20(5):537-41. doi: 10.1177/036354659202000509. PMID 1443321
- [Result] Cole BJ, Seroyer ST, Filardo G, Bajaj S, Fortier LA. Platelet-rich plasma: where are we now and where are we going? Sports Health. 2010 May;2(3):203-10. doi: 10.1177/1941738110366385. PMID 23015939
- [Result] Lopez-Vidriero E, Goulding KA, Simon DA, Sanchez M, Johnson DH. The use of platelet-rich plasma in arthroscopy and sports medicine: optimizing the healing environment. Arthroscopy. 2010 Feb;26(2):269-78. doi: 10.1016/j.arthro.2009.11.015. PMID 20141991
- [Result] Eppley BL, Woodell JE, Higgins J. Platelet quantification and growth factor analysis from platelet-rich plasma: implications for wound healing. Plast Reconstr Surg. 2004 Nov;114(6):1502-8. doi: 10.1097/01.prs.0000138251.07040.51. PMID 15509939
- [Result] Fufa D, Shealy B, Jacobson M, Kevy S, Murray MM. Activation of platelet-rich plasma using soluble type I collagen. J Oral Maxillofac Surg. 2008 Apr;66(4):684-90. doi: 10.1016/j.joms.2007.06.635. PMID 18355591
- [Result] Scordino LE, Deberardino TM. Biologic enhancement of meniscus repair. Clin Sports Med. 2012 Jan;31(1):91-100. doi: 10.1016/j.csm.2011.09.001. No abstract available. PMID 22108661
- [Result] Tumia NS, Johnstone AJ. Platelet derived growth factor-AB enhances knee meniscal cell activity in vitro. Knee. 2009 Jan;16(1):73-6. doi: 10.1016/j.knee.2008.08.008. Epub 2008 Oct 30. PMID 18976925
- [Result] Ishida K, Kuroda R, Miwa M, Tabata Y, Hokugo A, Kawamoto T, Sasaki K, Doita M, Kurosaka M. The regenerative effects of platelet-rich plasma on meniscal cells in vitro and its in vivo application with biodegradable gelatin hydrogel. Tissue Eng. 2007 May;13(5):1103-12. doi: 10.1089/ten.2006.0193. PMID 17348798
- [Result] de Vos RJ, Weir A, van Schie HT, Bierma-Zeinstra SM, Verhaar JA, Weinans H, Tol JL. Platelet-rich plasma injection for chronic Achilles tendinopathy: a randomized controlled trial. JAMA. 2010 Jan 13;303(2):144-9. doi: 10.1001/jama.2009.1986. PMID 20068208
- [Result] Benko A, Fraser-Hill M, Magner P, Capusten B, Barrett B, Myers A, Owen RJ; Canadian Association of Radiologists. Canadian Association of Radiologists: consensus guidelines for the prevention of contrast-induced nephropathy. Can Assoc Radiol J. 2007 Apr;58(2):79-87. PMID 17521052
- [Result] Kirkley A, Griffin S, Whelan D. The development and validation of a quality of life-measurement tool for patients with meniscal pathology: the Western Ontario Meniscal Evaluation Tool (WOMET). Clin J Sport Med. 2007 Sep;17(5):349-56. doi: 10.1097/JSM.0b013e31814c3e15. PMID 17873546